CLINICAL TRIAL: NCT06164327
Title: A Multicenter, Open Phase Ib Study of the Safety and Efficacy of BEBT-908 Combined With Drugs in the Treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Study of BEBT-908 Combined With Drugs in the Treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-908-P06
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Keywords: BEBT-908; Drug combination; Safety; Efficacy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — BEBT-908; Injections; Rituximab; Gemcitabine; Oxaliplatin; Etoposide; Ifosfamide; Carboplatin

STUDY DESIGN:
Intervention Model Description: The study sets up three cohorts of BEBT-908 combined with different drugs.The researchers decide whether to terminate the cohort study according to the safety and tolerability results of each cohort during the first cycle of medication. If the participants in the above three cohorts are unable to receive the treatment during the first cycle of medication, two alternative cohort studies will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BEBT-908 combined with R (Experimental): BEBT-908 for Injection,dosage of administration:22.5mg/m^2，frequency and duration of administration:on the 1st,3rd,5th,8th,10th and 12th days of each cycle in the 1st to 6th cycles,and 21 days as a cycle.
  Rituximab Injection,dosage of administration:375 mg/m^2,frequency and duration of administration:on the 1st day of each cycle, and 21 days as a cycle.
  Interventions: Drug: BEBT-908 for Injection; Drug: Rituximab Injection
- BEBT-908 combined with R-GemOx (Experimental): BEBT-908 for Injection,dosage of administration:15mg/m^2，frequency and duration of administration:on the 1st,3rd,5th,8th,10th and 12th days of each cycle in the 1st to 6th cycles,and 21 days as a cycle.
  Rituximab Injection,dosage of administration:375 mg/m^2,frequency and duration of administration:on the 1st day of each cycle in the 1st to 6th cycles, and 21 days as a cycle.
  Gemcitabine Hydrochloride for Injection，dosage of administration:1g/m^2,frequency and duration of administration:on the 2nd day of each cycle in the 1st to 6th cycles, and 21 days as a cycle.
  Oxaliplatin Injection,dosage of administration:100mg/m^2,frequency and duration of administration:on the 2nd day of each cycle in the 1st to 6th cycles, and 21 days as a cycle.
  Interventions: Drug: BEBT-908 for Injection; Drug: Rituximab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Oxaliplatin Injection
- BEBT-908 combined with R-ICE (Experimental): BEBT-908 for Injection,dosage of administration:15mg/m^2，frequency and duration of administration:on the 1st,3rd,5th,8th,10th and 12th days of each cycle in the 1st to 6th cycles,and 21 days as a cycle.
  Rituximab Injection,dosage of administration:375 mg/m^2,frequency and duration of administration:on the 1st day of each cycle in the 1st to 6th cycles, and 21 days as a cycle.
  Etoposide Injection,dosage of administration:100mg/m^2，frequency and duration of administration:on the 1st,2nd and 3rd days of each cycle in the 1st to 6th cycles,and 21 days as a cycle.
  Ifosfamide for Injection,dosage of administration:5000mg/m^2,frequency and duration of administration:on the 2nd day of each cycle in the 1st to 6th cycles, and 21 days as a cycle.
  Carboplatin Injection，dosage of administration:based on AUC=5, single dose ≤800 mg，frequency and duration of administration:on the 2nd day of each cycle in the 1st to 6th cycles, and 21 days as a cycle.
  Interventions: Drug: BEBT-908 for Injection; Drug: Rituximab Injection; Drug: Etoposide Injection; Drug: Ifosfamide for Injection; Drug: Carboplatin Injection
- BEBE-908 monotherapy (alternative cohort 1) (Experimental): BEBT-908 for Injection,dosage of administration:22.5mg/m^2，frequency and duration of administration:on the 1st,3rd,5th,8th,10th and 12th days of each cycle in the 1st to 6th cycles,and 21 days as a cycle.
  Interventions: Drug: BEBT-908 for Injection
- BEBT-908 combined with R-GemOx（alternative cohort 2） (Experimental): BEBT-908 for Injection,dosage of administration:22.5mg/m^2，frequency and duration of administration:on the 1st,3rd,5th,8th,10th and 12th days of each cycle in the 1st to 2nd cycles,and 21 days as a cycle.
  Rituximab Injection,dosage of administration:375 mg/m^2,frequency and duration of administration:on the 1st day of each cycle in the 3rd to 6th cycles, and 21 days as a cycle.
  Gemcitabine Hydrochloride for Injection，dosage of administration:1g/m^2,frequency and duration of administration:on the 2nd day of each cycle in the 3rd to 6th cycles, and 21 days as a cycle.
  Oxaliplatin Injection,dosage of administration:100mg/m^2,frequency and duration of administration:on the 2nd day of each cycle in the 3rd to 6th cycles, and 21 days as a cycle.
  Interventions: Drug: BEBT-908 for Injection; Drug: Rituximab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Oxaliplatin Injection

INTERVENTIONS:
Drug: BEBT-908 for Injection — BEBT-908 for Injection,dosage of administration:15mg/m^2 or 22.5mg/m^2，frequency and duration of administration:on the 1st,3rd,5th,8th,10th and 12th days of each cycle,and 21 days as a cycle.
  Other Names: CUDC-908
Drug: Rituximab Injection — Rituximab Injection,dosage of administration:375 mg/m^2,frequency and duration of administration:on the 1st day of each cycle, and 21 days as a cycle.
  Other Names: IDEC-C2B8
  Arms: BEBT-908 combined with R; BEBT-908 combined with R-GemOx; BEBT-908 combined with R-GemOx（alternative cohort 2）; BEBT-908 combined with R-ICE
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for Injection，dosage of administration:1g/m^2,frequency and duration of administration:on the 2nd day of each cycle, and 21 days as a cycle.
  Other Names: NSC 613327
  Arms: BEBT-908 combined with R-GemOx; BEBT-908 combined with R-GemOx（alternative cohort 2）
Drug: Oxaliplatin Injection — Oxaliplatin Injection，dosage of administration:100mg/m^2,frequency and duration of administration:on the 2nd day of each cycle, and 21 days as a cycle.
  Other Names: NSC 266046
  Arms: BEBT-908 combined with R-GemOx; BEBT-908 combined with R-GemOx（alternative cohort 2）
Drug: Etoposide Injection — Etoposide Injection,dosage of administration:100mg/m^2，frequency and duration of administration:on the 1st,2nd and 3rd days of each cycle,and 21 days as a cycle.
  Other Names: VP-16213
  Arms: BEBT-908 combined with R-ICE
Drug: Ifosfamide for Injection — Ifosfamide for Injection,dosage of administration:5000mg/m^2,24 hours of continuous intravenous drip，frequency and duration of administration:on the 2nd day of each cycle, and 21 days as a cycle.
  Other Names: NSC109724
  Arms: BEBT-908 combined with R-ICE
Drug: Carboplatin Injection — Carboplatin Injection，dosage of administration:based on AUC=5, single dose ≤800 mg，frequency and duration of administration:on the 2nd day of each cycle, and 21 days as a cycle.
  Other Names: NSC 241240
  Arms: BEBT-908 combined with R-ICE

SUMMARY:
This is a multicenter, open Phase Ib clinical study to evaluate the safety,efficacy and pharmacokinetics of BEBT-908 combined with Rituximab (R) or combined with Rituximab-Gemcitabine-Oxaliplatin (R-GemOx) or combined with Rituximab-Ifosfamide-Carboplatin-Etoposide (R-ICE) in the treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL).

DETAILED DESCRIPTION:
This study sets up three cohorts, including BEBT-908 combined with R, BEBT-908 combined with R-ICE, and BEBT-908 combined with R-GemOx. The researchers decide whether to terminate the cohort study according to the safety and tolerability results of each cohort during the first cycle of medication. If the participants in the above three cohorts are unable to receive the treatment during the first cycle of medication, two alternative cohort studies will be conducted. Namely, BEBT-908 monotherapy (alternative cohort 1), adjustment of BEBT-908 combined with GemOx administration regimen (alternative cohort 2).

The study process for each participant includes a screening period, a treatment period, and a post-treatment follow-up period. During treatment, participants are evaluated for tumors every 6 weeks, follow up after termination of treatment with efficacy follow-up every 6 weeks for those without disease progression and survival follow-up every 3 months until disease progression (PD), death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurred first).

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing to sign the informed consent form (ICF) after comprehensive understanding;
2. Age ≥18 years and ≤75 years, both male and female;
3. The pathology was confirmed as diffuse large B-cell lymphoma according to the 2016 World Health Organization classification definition;
4. Evaluation by Positron Emission Computed Tomography (PET-CT) or Computed Tomography (CT) or Magnetic resonance imaging (MRI) using Lugano 2014 standard, with measurable lesion injection;
5. Must have recurrent or refractory diffuse large B-cell lymphoma after at least 1 systemic therapy, and at least 1 systemic therapy included CD20 antibody;
6. Eastern Cooperative Oncology Group (ECOG) scores 0-2 points;
7. Life expectancy >12 weeks;
8. The level of organ function must meet the following requirements:

Peripheral blood:

1. Absolute neutrophil count (ANC) ≥1000/μL;
2. Hemoglobin (HGB) ≥8g/dL;
3. Platelet count (PLT) ≥100,000/μL;

Liver function:

1. Serum total bilirubin ≤1.5×ULN (for patients with Gilbert syndrome, total bilirubin <3.0×ULN and Direct bilirubin within normal range);
2. Serum creatinine <1.5×ULN;
3. ALT, AST or ALP≤2.5×ULN (≤5×ULN when liver involvement occurs).

Exclusion Criteria:

1. Known severe allergy to the investigational drug or any of its excipients;
2. Due to the possibility of genotoxicity, mutagenicity and teratogenicity of the investigational drug, the following subjects should be excluded:

   1. Men and women who have not had sperm or egg preservation in vitro before the trial and plan to have another child within 5 years unless subsequent studies confirm reproductive safety;
   2. Pregnant or lactating women;
3. Primary central nervous system lymphoma or lymphoma invading the central nervous system;
4. Previous chronic lymphoma transformation (such as Richter syndrome, prelymphocytic leukemia, etc.);
5. There are other active malignant tumors requiring treatment that may interfere with the study;
6. Pre-trial treatment:

   1. Received any persistent or intermittent PI3K inhibitor and HDAC inhibitor prior to enrollment or received other small-molecule targeted drug therapy within 2 weeks;
   2. Received BEBT-908 (not allowed to be in all cohorts) or R-ICE (not allowed to be in cohorts with BEBT-908+R-ICE) or R-GemOx (not allowed to be in cohorts with BEBT-908+R-GemOx) prior to enrollment;
   3. Autologous hematopoietic stem cell transplantation within 3 months before enrollment;
   4. Received radiotherapy that affected the evaluation of the efficacy of the study or local supportive radiotherapy that affected the bone marrow function of the subjects within 3 months before enrollment;
   5. Received myelosuppressive chemotherapy or biotherapy within 3 weeks prior to enrollment;
   6. Used Chinese medicines and proprietary Chinese medicines with anti-tumor effects within 2 weeks before enrollment;
   7. Undergone major surgery other than tumor biopsy within 4 weeks prior to enrollment, or the side effects of surgery had not stabilized;
   8. Any hematopoietic colony-stimulating factor (e.g., granulocyte colony-stimulating factor G-CSF, granulocyte macrophage colony-stimulating factor GM-CSF) or thrombopoietin TPO were treated within 2 weeks prior to enrollment；
   9. Received prednisone >10mg daily (or another equivalent dose of glucocorticoid) within 7 days prior to enrollment;
   10. Received chimeric antigen receptor T cell immunotherapy (CAR-T therapy) within 3 months before enrollment;
7. Persistent grade 2 or higher [Common Terminology Criteria for Adverse Events V5.0 standard (CTCAE V5.0 standard)] toxicity after previous treatment (chemotherapy or biotherapy), not stable at enrollment (except alopecia);
8. Active clinical severe infection of grade 2 or above (CTCAE V5.0 standard);
9. Complicated diseases:

   1. diabetes mellitus with poor glycemic control (random glycemic value ≥11.1mmol/L after hypoglycemic treatment, or glycosylated hemoglobin（HbA1c）≥ 8.5%);
   2. severe lung disease (CTCAE V5.0 grade III-IV);
   3. Serious heart disease;
   4. have significant kidney or liver dysfunction;
   5. Poorly controlled active diseases such as hepatitis B or C;
   6. Known human immunodeficiency virus (HIV) positive;
   7. A history of mental illness, family history of mental illness, or mood disorder, as judged by the investigator or psychologist, and the researcher judged that they were not suitable for inclusion;
   8. Combination of anticoagulation and antiplatelet therapy is required during the study period;
   9. uncontrolled hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg);
   10. Serious physical disease combined with the risk of major bleeding or a history of major bleeding;
10. Combined with use of drugs that cause QT interval prolongation or torsional ventricular tachycardia;
11. Receiving cytochrome P450 (CYP) 3A4 isozyme suppressant or strongly induced drug therapy during the first 4 weeks of enrollment；
12. Participated in other clinical trials and used investigational drugs within 4 weeks before enrollment;
13. Any condition that the investigator determines to be unstable or likely to compromise the subject's safety and compliance with the study;
14. Subjects deemed unsuitable for treatment with this protocol by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
ORR | Every 6 weeks，assessed up to 24 months.
  Objective response rate
AE | From the first administration of the study drug to 28 days after the last administration of the study drug
  Adverse event

SECONDARY OUTCOMES:
ORR-EoT | Every 6 weeks，assessed up to 6 treatment cycles (each cycle is 21 days).
  Objective response rate after completion of treatment
PFS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival
OS | From date of administration until date of death from any cause, assessed up to 24 months.
  Overall Survival
CBR | Every 6 weeks，assessed up to 24 months.
  Clinical benefit rate
DOR | Every 6 weeks，assessed up to 24 months.
  Duration of Response
DCR | Every 6 weeks，assessed up to 24 months.
  Disease Control Rate
TTR | Every 6 weeks，assessed up to 24 months.
  Treatment response time
Tmax | From 1 hour before dosing on day 1 and day 12 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 8 and day 10 of the first cycle (each cycle is 21 days).
  Time of peak Plasma Concentration
Cmax | From 1 hour before dosing on day 1 and day 12 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 8 and day 10 of the first cycle (each cycle is 21 days).
  Peak Plasma Concentration
t1/2 | From 1 hour before dosing on day 1 and day 12 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 8 and day 10 of the first cycle (each cycle is 21 days).
  Half-life of plasma drug concentrations
AUC0-t | From 1 hour before dosing on day 1 and day 12 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 8 and day 10 of the first cycle (each cycle is 21 days).
  Area under the plasma concentration time curve from 0 hour to last time of quantifiable concentration after administration
CL | From 1 hour before dosing on day 1 and day 12 of the first cycle to 48 hours after dosing, and from 1 hour before dosing on day 8 and day 10 of the first cycle (each cycle is 21 days).
  apparent plasma clearance

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Phd, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China